CLINICAL TRIAL: NCT02458339
Title: Phase I Study of Methotrexate Infusion Into the Fourth Ventricle in Children With Recurrent Malignant Fourth Ventricular Brain Tumors
Brief Title: Methotrexate Infusion Into Fourth Ventricle in Children With Recurrent Malignant Fourth Ventricular Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, David Ilan Sandberg, Director of Pediatric Neurosurgery, Associate Professor, Departments of Pediatric Surgery and Neurosurgery UTHealth Medical School, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0035
Record Dates: First submitted 2015-05-20; First posted 2015-06-01 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Brain Tumor, Recurrent; Malignant Neoplasm of Fourth Ventricle of Brain
Keywords: Brain tumor; Malignant Fourth Ventricular Brain Tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): 3 consecutive cycles of intraventricular methotrexate infusions into implanted fourth ventricle catheter/Ommaya reservoir following surgical catheter placement into fourth ventricle, each cycle will be of 4 weeks duration. During the first 3 weeks, methotrexate will be infused twice weekly on days 1 and 4 (+/- 2 days). The 4th week is a rest week.
  Interventions: Procedure: Ommaya Reservoir; Drug: Methotrexate

INTERVENTIONS:
Procedure: Ommaya Reservoir — Surgical catheter placement into the fourth ventricle of the brain
Drug: Methotrexate — 4, 6, or 8 mg into fourth ventricle of the brain via the Ommaya Reservoir for 2 days a week for 3 weeks with week 4 is a rest week. Each patient will undergo three cycles.

SUMMARY:
The goal of this clinical research study is to establish the maximum tolerated dose (MTD) of direct administration of methotrexate into the fourth ventricle of the brain in patients with recurrent malignant brain tumors including medulloblastoma, primitive neuroectodermal tumors (PNET), atypical teratoid/rhabdoid tumors (AT/RT), and ependymoma.

Methotrexate is designed to block cancer cells from dividing, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

DETAILED DESCRIPTION:
If the participant is eligible to take part in this study, the participant will have surgery to place a catheter into the ommaya reservoir. The ommaya reservoir is a catheter system that allows drugs to be administered directly to parts of the brain. This catheter will be used for the infusion of methotrexate directly into the 4th ventricle of the brain, which is 1 of the 4 connected fluid-filled cavities in the brain.

If the study doctor thinks it is necessary, based on the location of the tumor, the tumor may also be removed while the participant is already under anesthesia just before the catheter is placed.

Study Drug Administration:

The participant will receive 3 cycles of intraventricular methotrexate into the fourth ventricle. Each cycle will be of 4 weeks duration. During the first 3 weeks (Day 1-7 weekly) methotrexate will be infused twice weekly on days 1 and 4 (+/-2 days). The 4th week will be a rest week.

Methotrexate will be infused through the ommaya reservoir catheter directly into the 4th ventricle of the brain starting at a minimum of 7 days after the catheter placement surgery. A MRI will be done to confirm adequate cerebrospinal fluid flow. The infusion should last about 3 minutes each time.

If the participant already has an ommaya catheter, methotrexate will begin after an MRI has confirmed adequate cerebrospinal fluid flow.

Study Visits:

Prior to Cycle 1:

* Medical history will be reviewed and any updates to health will be recorded
* A physical with vital signs and neurological exam will be done.
* Blood (about 1 teaspoon) will be drawn for routine test
* A MRI scan of the brain and spine will be done to check the status of the disease.

On the days of Methotrexate Infusion:

* A physical with vital signs and neurological exam will be done
* A Ommaya reservoir tap (a catheter is placed into the Ommaya reservoir to give the methotrexate infusion).
* Cerebrospinal fluid (about 1 teaspoon) will be collected for routine tests.

Within 7 days of completing Cycle 3:

* A physical with vital signs and neurological exam will be done.
* A lumbar puncture will be done.
* A MRI scan of the brain and spine will be done to check the status of the disease.

Length of Study:

The participant will receive up to 3 cycles of the methotrexate, as long as the doctor thinks it is in their best interest. The participant will no longer be able to receive the study drug if the disease gets worse, if intolerable side effects occur, or if unable to follow study directions.

This is an investigational study. Methotrexate is FDA approved and commercially available for infusion directly into brain tumors. The infusion of methotrexate into the 4th ventricle of the brain is investigational,

Up to 18 patients will be enrolled in this study. All will be enrolled at Children's Memorial Hermann Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Patients with histologically verified medulloblastoma, primitive neuroectodermal tumor (PNET), atypical teratoid/rhabdoid tumor (AT/RT), ependymoma, or choroid plexus carcinoma with recurrence or progression involving the brain and /or spine. Patients with these tumors who did not present at diagnosis in the posterior fossa but have relapsed in the posterior fossa will be eligible. Patients who initially presented with disease in the posterior fossa but have now relapsed outside the posterior fossa will also be eligible.
2. Patient must have either measurable or evaluable tumor as assessed by MRI of the brain and total spine.
3. An implanted catheter in the fourth ventricle attached to an Ommaya reservoir or agreement to have one placed.
4. A minimum of 7 days between last dose of systemic chemotherapy and/or radiation therapy and first infusion of methotrexate into fourth ventricle.
5. Life expectancy of at least 12 weeks in the opinion of the PI.
6. Lansky score of 50 or greater if ≤16 years of age or Karnofsky score of 50 or greater if > 16 years of age.
7. Existing neurological deficits such as weakness, gait instability, cranial nerve deficits, or any other problems caused by the patient's disease or previous treatments must have been stable for a minimum of 1 week prior to study enrollment.
8. Patients must have recovered from the acute toxic effects of all prior anticancer chemotherapy.
9. Adequate bone marrow function defined by peripheral absolute neutrophil count (ANC) ≥ 500/ µL, platelet count ≥ 50,000/ µL(transfusion independent), and hemoglobin ≥ 9.0 gm/dL (may receive RBC transfusions)
10. Patient or patient's legal representative, parent (s), or guardian able to provide written informed consent.

Exclusion Criteria:

1. Enrolled in another treatment protocol
2. Has received another investigational or chemotherapy agent or radiation therapy with in 7 days prior to methotrexate infusion into the fourth ventricle
3. Evidence of untreated infection
4. Pregnant or lactating women

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of the direct administration of methotrexate into the fourth ventricle of the brain as determined by NCI's CTCAE | 3 months
  Maximum Tolerated Dose (MTD) is determined using the criteria established by the National Cancer Institute's (NCI's) Common Terminology Criteria for Adverse Events V4.0 (CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: David I Sandberg, MD, Principal Investigator — UTHealth Medical School
Locations (1):
- UTHealth & Children's Memorial Hermann Hospital, Houston, Texas, United States